CLINICAL TRIAL: NCT03049540
Title: Effect of Phosphodiesterase-5 Inhibition With Tadalafil on SystEmic Right VEntricular Size and Function - a Multi-center, Double-blind, Randomized, Placebo-controlled Clinical Trial - SERVE Trial
Brief Title: Effect of Phosphodiesterase-5 Inhibition With Tadalafil on SystEmic Right VEntricular Size and Function
Acronym: SERVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: V1 2016-10-12
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Heart Defects, Congenital; Transposition of Great Vessels With Ventricular Inversion
MeSH Terms: conditions — Heart Defects, Congenital; Congenitally Corrected Transposition of the Great Arteries | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil (Active Comparator): Tadalafil 20 MG, p.o., once per day for 3 years
  Interventions: Drug: Tadalafil 20 MG
- Placebo (Placebo Comparator): Placebo 20 MG, p.o., once per day for 3 years
  Interventions: Drug: Placebo 20 MG

INTERVENTIONS:
Drug: Tadalafil 20 MG — Multi-center, double-blind, 1:1 randomized, placebo-controlled clinical trial with Tadalafil
  Arms: Tadalafil
Drug: Placebo 20 MG — Multi-center, double-blind, 1:1 randomized, placebo-controlled clinical trial with Tadalafil
  Arms: Placebo

SUMMARY:
This study assesses in a double-blind, randomized, placebo-controlled multi-center pilot trial the effect of PDE-5 inhibition with Tadalafil on right ventricle size and function, exercise capacity and neurohumoral activation in adults with congenital heart disease and a right ventricle in subaortic position over a 3-year follow-up period.

DETAILED DESCRIPTION:
Currently, there are an estimated 300-600 adults living in Switzerland with congenital heart disease (CHD) and a right ventricle (RV) in subaortic (systemic) position. This includes adults with prior atrial switch operations for complete transposition of the great arteries (D-TGA) and adults with congenitally corrected transposition of the great arteries (ccTGA). Although midterm survival is favourable, late outcome is compromised by ventricular dysfunction of the systemic RV, end-stage heart failure, and premature death. Medical heart failure therapy (ACE-inhibitors, beta-blockers, aldosterone antagonists) has been shown to improve ventricular function and survival in patients with left heart failure from acquired heart disease. Unfortunately, case-reports and studies failed to show similar clinical benefits of these drugs in adults with a failing systemic RV. Currently, the only established end-stage therapy for a failing systemic RV is heart transplantation. Given the ubiquitous shortage of donor organs and the number of adults at risk, medical options to improve the fate of patients with a systemic RV are urgently needed.

The RV and left ventricle (LV) have different embryological origins, myocardial architecture and contractile properties. In response to increased afterload, as in an RV in systemic position, the RV expresses a fetal gene pattern, with an increase in phosphodiesterase (PDE)-5 expression. PDE-5 is not expressed in the normal RV, but is up-regulated in the hypertrophied RV. PDE-5 inhibition increases contractility in experimental models of RV hypertrophy, but not in the normal RV. In clinical practice, the effects of PDE-5 inhibition on systemic RV function and exercise capacity in adults with TGA have not been tested.

This study assesses in a double-blind, randomized, placebo-controlled multi-center pilot trial the effect of PDE-5 inhibition with Tadalafil on RV size and function, exercise capacity and neurohumoral activation in adults with a systemic RV over a 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Systemic right ventricle due to prior atrial switch operations for complete transposition of the great arteries (D-TGA) due to congenitally corrected transposition of the great arteries (ccTGA).

Exclusion Criteria:

* Incapability of giving informed consent
* Myocardial infarction, stroke, or open heart surgery within the 3 months prior to baseline visit
* Expected heart transplant within the next 6 months starting from baseline
* Pregnant or nursing women (a pregnancy test is mandatory prior to randomization; women of childbearing potential must agree to use reliable contraception from randomization to end of study treatment)
* Severe renal insufficiency (Creatinine clearance ≤ 30 ml/min)
* Severe hepatic insufficiency (Child-Pugh-Class C)
* Hypotension with blood pressures < 90/50 mmHg at the baseline visit
* Hypersensibility to Tadalafil
* Allergy to iodinated (in patients undergoing CMDCT) or Gadolinium-based (in patients undergoing CMR) contrast agents.
* Co-medication with nitrates
* Regular use of "poppers", i.e. alkyl nitrites, that are inhaled for recreational purposes, including as club drugs used at dance clubs.
* Co-medication with potent CYP3A4 inhibitors: Ketoconazole, Ritonavir, Rifampicin
* Co-medication with other PDE-5 inhibitors for erectile dysfunction during the last four weeks prior to baseline visit
* Medical history of Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION)
* Hereditary Galactose intolerance, Lactase deficiency or Glucose-Galactose-Malabsorption
* Participation at another clinical trial in which the primary endpoint has not been reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Systemic right ventricle endsystolic volume | 3 years
  Assess of the improvement of Tadalafil on systemic right ventricle endsystolic volume measured by cardiovascular magnetic resonance imaging (CMR) or cardiac multirow detector computed tomography (CMDCT) in patients with contraindications for cardiac MRI

SECONDARY OUTCOMES:
Systemic right ventricle ejection fraction | 3 years
  Systemic right ventricle ejection fraction measured by CMR or CMDCT
Cardiopulmonary exercise capacity | 3 years
  Assess the effects of PDE-5 inhibition on cardiopulmonary exercise capacity
Serum neurohormonal activation | 3 years
  Assess the effects of PDE-5 inhibition on serum neurohormonal activation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schwerzmann, MD, Principal Investigator — Bern University Hospital, Zentrum fuer angeborene Herzfehler
Locations (7):
- Universitätsklinik für Innere Medizin II, Medizinische Universität Wien, Vienna, Austria
- Switzerland (6):
  - Kardiologie Universitätsspital Basel, Basel
  - Bern University Hospital, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Universitäres Herzzentrum, Zurich

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Roos-Hesselink JW, Meijboom FJ, Spitaels SE, van Domburg R, van Rijen EH, Utens EM, McGhie J, Bos E, Bogers AJ, Simoons ML. Decline in ventricular function and clinical condition after Mustard repair for transposition of the great arteries (a prospective study of 22-29 years). Eur Heart J. 2004 Jul;25(14):1264-70. doi: 10.1016/j.ehj.2004.03.009. PMID 15246646
- [Result] van der Bom T, Bouma BJ, Meijboom FJ, Zwinderman AH, Mulder BJ. The prevalence of adult congenital heart disease, results from a systematic review and evidence based calculation. Am Heart J. 2012 Oct;164(4):568-75. doi: 10.1016/j.ahj.2012.07.023. PMID 23067916
- [Result] Marelli AJ, Mackie AS, Ionescu-Ittu R, Rahme E, Pilote L. Congenital heart disease in the general population: changing prevalence and age distribution. Circulation. 2007 Jan 16;115(2):163-72. doi: 10.1161/CIRCULATIONAHA.106.627224. Epub 2007 Jan 8. PMID 17210844
- [Result] Mylotte D, Pilote L, Ionescu-Ittu R, Abrahamowicz M, Khairy P, Therrien J, Mackie AS, Marelli A. Specialized adult congenital heart disease care: the impact of policy on mortality. Circulation. 2014 May 6;129(18):1804-12. doi: 10.1161/CIRCULATIONAHA.113.005817. Epub 2014 Mar 3. PMID 24589851
- [Result] Cuypers JA, Eindhoven JA, Slager MA, Opic P, Utens EM, Helbing WA, Witsenburg M, van den Bosch AE, Ouhlous M, van Domburg RT, Rizopoulos D, Meijboom FJ, Bogers AJ, Roos-Hesselink JW. The natural and unnatural history of the Mustard procedure: long-term outcome up to 40 years. Eur Heart J. 2014 Jul 1;35(25):1666-74. doi: 10.1093/eurheartj/ehu102. Epub 2014 Mar 18. PMID 24644309
- [Result] Vejlstrup N, Sorensen K, Mattsson E, Thilen U, Kvidal P, Johansson B, Iversen K, Sondergaard L, Dellborg M, Eriksson P. Long-Term Outcome of Mustard/Senning Correction for Transposition of the Great Arteries in Sweden and Denmark. Circulation. 2015 Aug 25;132(8):633-8. doi: 10.1161/CIRCULATIONAHA.114.010770. Epub 2015 Jul 16. PMID 26185211
- [Result] Roche SL, Redington AN. The failing right ventricle in congenital heart disease. Can J Cardiol. 2013 Jul;29(7):768-78. doi: 10.1016/j.cjca.2013.04.018. PMID 23790549
- [Result] van der Bom T, Winter MM, Bouma BJ, Groenink M, Vliegen HW, Pieper PG, van Dijk AP, Sieswerda GT, Roos-Hesselink JW, Zwinderman AH, Mulder BJ. Effect of valsartan on systemic right ventricular function: a double-blind, randomized, placebo-controlled pilot trial. Circulation. 2013 Jan 22;127(3):322-30. doi: 10.1161/CIRCULATIONAHA.112.135392. Epub 2012 Dec 17. PMID 23247302
- [Result] Dos L, Pujadas S, Estruch M, Mas A, Ferreira-Gonzalez I, Pijuan A, Serra R, Ordonez-Llanos J, Subirana M, Pons-Llado G, Marsal JR, Garcia-Dorado D, Casaldaliga J. Eplerenone in systemic right ventricle: double blind randomized clinical trial. The evedes study. Int J Cardiol. 2013 Oct 15;168(6):5167-73. doi: 10.1016/j.ijcard.2013.07.163. Epub 2013 Jul 25. PMID 23972966
- [Result] Nagendran J, Archer SL, Soliman D, Gurtu V, Moudgil R, Haromy A, St Aubin C, Webster L, Rebeyka IM, Ross DB, Light PE, Dyck JR, Michelakis ED. Phosphodiesterase type 5 is highly expressed in the hypertrophied human right ventricle, and acute inhibition of phosphodiesterase type 5 improves contractility. Circulation. 2007 Jul 17;116(3):238-48. doi: 10.1161/CIRCULATIONAHA.106.655266. Epub 2007 Jul 2. PMID 17606845
- [Result] Schwartz BG, Levine LA, Comstock G, Stecher VJ, Kloner RA. Cardiac uses of phosphodiesterase-5 inhibitors. J Am Coll Cardiol. 2012 Jan 3;59(1):9-15. doi: 10.1016/j.jacc.2011.07.051. PMID 22192662
- [Result] Kloner RA, Jackson G, Hutter AM, Mittleman MA, Chan M, Warner MR, Costigan TM, Vail GM. Cardiovascular safety update of Tadalafil: retrospective analysis of data from placebo-controlled and open-label clinical trials of Tadalafil with as needed, three times-per-week or once-a-day dosing. Am J Cardiol. 2006 Jun 15;97(12):1778-84. doi: 10.1016/j.amjcard.2005.12.073. Epub 2006 Apr 27. PMID 16765134
- [Result] Greutmann M, Tobler D, Engel R, Heg D, Mueller C, Frenk A, Gabriel H, Rutz T, Buechel RR, Willhelm M, Trachsel L, Freese M, Ruperti-Repilado FJ, Valsangiacomo Buechel E, Beitzke D, Haaf P, Wustmann K, Schwitz F, Possner M, Schwitter J, Bouchardy J, Schwerzmann M; SERVE Investigators. Effect of phosphodiesterase-5 inhibition on SystEmic Right VEntricular size and function. A multicentre, double-blind, randomized, placebo-controlled trial: SERVE. Eur J Heart Fail. 2023 Jul;25(7):1105-1114. doi: 10.1002/ejhf.2924. Epub 2023 Jun 13. PMID 37264734
- [Result] Tobler D, Bouchardy J, Reto E, Heg D, Muller C, Frenk A, Gabriel H, Schwitter J, Rutz T, Buechel RR, Willhelm M, Trachsel L, Freese M, Greutmann M, Schwerzmann M; SERVE trial. Effect of phosphodiesterase-5 inhibition with Tadalafil on SystEmic Right VEntricular size and function - A multi-center, double-blind, randomized, placebo-controlled clinical trial - SERVE trial - Rational and design. Int J Cardiol. 2017 Sep 15;243:354-359. doi: 10.1016/j.ijcard.2017.05.079. Epub 2017 May 23. PMID 28566262
- [Derived] Castiglione A, Schwerzmann M, Bouchardy J, Buechel RR, Engel R, Freese M, Gabriel H, Greutmann M, Heg D, Mueller C, Possner M, Ruperti-Repilado FJ, Rutz T, Schwitter J, Thomet C, Tobler D, Wilhelm M, Wustmann K, Schwitz F; SERVE trial. Stable Longitudinal Quality of Life in the SERVE Trial Among Adults With Transposition of the Great Arteries and a Systemic Right Ventricle. CJC Pediatr Congenit Heart Dis. 2024 Dec 12;4(2):81-91. doi: 10.1016/j.cjcpc.2024.12.001. eCollection 2025 Apr. PMID 40470125
- [Derived] Ruperti-Repilado FJ, Tran F, Haaf P, Lopez-Ayala P, Greutmann M, Schwerzmann M, Bouchardy J, Gabriel H, Stambach D, Rutz T, Schwitter J, Wustmann K, Freese M, Mueller C, Tobler D. Prognostic Value and Determinants of High-Sensitivity Cardiac Troponin T in Patients With a Systemic Right Ventricle: Insights From the SERVE Trial. J Am Heart Assoc. 2024 May 21;13(10):e034776. doi: 10.1161/JAHA.123.034776. Epub 2024 May 10. PMID 38726920